CLINICAL TRIAL: NCT04556994
Title: Comparison of Phase 1 Cardiac Rehabilitation With and Without Lower Limb Paddling Effects in Post CABG Patients.
Brief Title: Phase 1 Cardiac Rehabilitation With and Without Lower Limb Paddling Effects in Post CABG Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/00699 Muhammad Faizan
Record Dates: First submitted 2020-09-16; First posted 2020-09-21 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Cardiac Rehabilitation; CABG; Ergometer
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1 Cardiac Rehabilitation (Active Comparator): Phase 1 Cardiac Rehabilitation
  Interventions: Other: Phase 1 Cardiac Rehabilitation
- Phase 1 Cardiac Rehabilitation with Lower Limb Paddling (Experimental): Phase 1 Cardiac Rehabilitation with lower limb paddling
  Interventions: Other: Phase 1 Cardiac Rehabilitation with Lower Limb Paddling

INTERVENTIONS:
Other: Phase 1 Cardiac Rehabilitation — Step 1:Breathing exercises, 3 sets of 10 repetitions. Active upper and lower extremity exercises, 3 sets of 10 repetitions; bed inclined at 45°.
  Step 2:Active exercises as in step 1. Stay in the upright position and perform walking on the spot for three series of 1 min.
  Step 3:Active exercises as in step 2. Ambulation within the inpatient wards (7 min). Transfer to an allocated chair beside the bed (at least 30 min).
  Step 4:Same exercises as in step 3. Ambulation within the inpatient wards (10 min). Transfer to an allocated chair beside the bed (at least 1 h).
  Step 5:Same exercises as in step 4. Ambulation within the inpatient wards (15 min). Transfer to an allocated chair beside the bed (at least 2 h).
  Step 6:Active exercises from the previous day. Ambulation within the inpatient wards (20 min). Step training (3 times continuously, 20 cm standardized step).
  Step 7:Exercises from the previous day. Step training (6 times continuously, 20 cm standardized step).
  Arms: Phase 1 Cardiac Rehabilitation
Other: Phase 1 Cardiac Rehabilitation with Lower Limb Paddling — Step 1 to step 6 of Phase 1 Cardiac Rehabilitation given to the patients along with Lower limb exercise on Paddler lasting 20 min (5-min warm-up, 10 min of low-intensity exercise, and 5-min recovery), 30 rpm ( rotation per minute)
  Arms: Phase 1 Cardiac Rehabilitation with Lower Limb Paddling

SUMMARY:
To compare the effect of Phase 1 cardiac rehabilitation with lower limb paddling, with phase 1 cardiac rehabilitation without lower limb paddling Effects in Post Coronary artery bypass graft (CABG) Patients.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) is the most common type of heart disease. CAD happens when the arteries that supply blood to heart muscle become hardened and narrowed. This is due to the buildup of cholesterol and other material, called plaque, on their inner walls. This buildup is called atherosclerosis. As it grows, less blood can flow through the arteries. As a result, the heart muscle can't get the blood or oxygen it needs. This can lead to chest pain (angina) or a heart attack. Most heart attacks happen when a blood clot suddenly cuts off the hearts' blood supply, causing permanent heart damage.

Previous studies reported positive effects of early exercise in the ICU on these measures . In a meta-analysis published earlier, early mobilization increased the number of ventilator-free days during hospitalization, but not the duration of Minute ventilation (MV). A possible explanation is that many patients without MV were included . As a result, these results should be interpreted with caution. The mortality rate is a traditional measure of the health status of critically ill patients. Muscle weakness is associated with increased mortality. Physical therapy in the intensive care unit (ICU) had no effect on mortality in many previous systematic reviews and meta-analyses. Similar to previous studies, early mobilization did not improve ICU mortality, hospital mortality, or 28-day mortality rates in the previously published meta-analysis. The discharged-to-home rate is an important prognostic indicator for critically ill patients, first showed that early mobilization increased the discharged-to-home rate compared to the control group.

In previous study it was concluded that, after the performance of the mobilization protocol, the patients in the Immunoglobulins (IG) improved the distance walked in the 6 min walk test (6MWT), which was assessed during 7 postoperative days and 60 days after hospital discharge, and it was less time in ICU and lower prevalence of pulmonary complications, when compared to the control group (CG). It was also concluded that with the results obtained from their study, it was possible to introduce an early mobilization protocol in the ICU routinely unit and sensitize the medical board about the importance of proper physiotherapy conduct.

Another previously conducted study states that regardless of the different techniques and periods of mobilization applied, early mobilization may be initiated safely in the ICU setting and appears to decrease the incidence of Intensive care unit-acquired weakness (ICU-AW), improve the functional capacity, and increase the number of patients who are able to stand, number of ventilator-free days and discharged-to-home rate without increasing the rate of adverse events. However, due to the substantial heterogeneity among the included studies, the evidence has a low quality.

Previous study states the importance of this approach; this has been emphasized in previous studies on experienced paddlers, rowers, cross-country skiers, cyclists and runners. However, some studies in sports that depend upon a high lower extremity documented a dependence of results from a specific Paddler on the season when the test was undertaken. During paddling, ventilatory functions are also very important. Values for the maximal minute ventilation (Vmax) and tidal volume obtained in the cycle ergometer were higher than in paddling in previous studies. During endurance performance the tidal volume depends on age, sex and constitutional factors and, in athletes, mainly on the nature and duration.The Max oxygen consumption (VO2) differences between maximal cycling and paddling were non-significant in previous studies. The ventilation equivalent affords insight into the economy of respiration. The magnitude is dependent on constitutional factors, especially on morphological conditions of the respiratory system, and partly on sex, age and, especially in athletes, on the economy of ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 20 and 30 kg/m2
* Hemodynamic stability with or without use of positive inotropic drugs
* Absence of arrhythmias and angina
* Mean blood pressure (MBP) 60 ⩽ MBP ⩽ 100 mmHg
* Heart rate (HR) 60 ⩽ HR ⩽ 100 bpm without respiratory distress
* Respiratory rate (RR) ⩽ 20 without signs of infection

Exclusion Criteria:

* Previous pulmonary disease and acute lung disease
* Mechanical ventilation >24 h
* Left ventricular ejection fraction (LVEF) <35% or >54%
* Surgical reintervention
* Intraoperative death or any contraindications for the proposed measurements and/or treatment
* Contraindications for the 6MWT or any proposed protocol
* Orthopedic impairments
* Unstable angina
* HR >120 bpm at rest, and systolic blood pressure >180 mmHg or diastolic >100 mmHg.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Functional independence | 1 week
  The Functional Independence Measure (FIM) is an 18-item measurement tool that explores an individual's physical, psychological and social function. The tool is used to assess a patient's level of disability as well as change in patient status in response to rehabilitation or medical intervention.
  The higher the score is for a task, the more independent a person is at performing the task. For example, a score of 1 indicates that a person needs total assistance with a task, while a score of 7 means a person can perform a task with complete independence.
Self-efficacy Formative Questionnaire | 1 week
  The Self-Efficacy Formative Questionnaire was developed in 2015 by Research Collaboration. An extensive review of related research resulted in identifying the two components essential for developing self-efficacy. Positive self-efficacy increased when students both believe that ability can grow with effort, as well as believed in their abilities to meet specific goals. The questionnaire was tested for reliability using Cronbach's coefficient alpha2
  Results are displayed on a 100-point scale. These scores can be interpreted similar to grades (e.g., 70-79 is a C)
Arterial blood gases (Ph) | 1 week
  An arterial blood gas (ABG) test measures the acidity (pH) and the levels of oxygen and carbon dioxide in the blood from an artery. This test is used to check how well your lungs are able to move oxygen into the blood and remove carbon dioxide from the blood.
  Normal blood pH ranges from 7.35 to 7.45 this is slightly to the alkaline side of the scale. If the pH is at the low end of the scale or if it is actually below 7.35, the condition is acidemia. Thus if it above 7.45 it is described as alkalemia.
Ejection fraction | 1 week
  Echocardiography is a test that uses sound waves to produce live images of your heart. The image is an echocardiogram. This test allows your doctor to monitor how your heart and its valves are functioning. Ejection fraction is a measurement of the percentage of blood leaving your heart each time it contracts. The heart contracts and relaxes.
  A normal heart's ejection fraction may be between 50 and 70 percent. A ejection fraction measurement under 40 percent may be evidence of heart failure or cardiomyopathy.
  EF from 41 to 49 percent may be considered "borderline." It does not always indicate that a person is developing heart failure. Instead, it may indicate damage, perhaps from a previous heart attack.
  An ejection fraction measurement higher than 75 percent may indicate a heart condition such as hypertrophic cardiomyopathy.
Quality of Life SF-36 questionnaire | 1 week
  The Short Form 36 Health Survey Questionnaire (SF-36) questionnaire consists of eight scales yielding two summary measures: physical and mental health. The physical health measure includes four scales of physical functioning (10 items), role-physical (4 items), bodily pain (2 items), and general health (5 items). The mental health measure is composed of vitality (4 items), social functioning (2 items), role-emotional (3 items), and mental health (5 items). A final item, termed self-reported health transition, is answered by the client but is not included in the scoring process.
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.

CONTACTS AND LOCATIONS:
Overall Officials: Iqbal Tariq, MsCPPT, Principal Investigator — Riphah International University
Locations (1):
- Rawal General & Dental Hospital, Islamabad, Fedral, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Busch JC, Lillou D, Wittig G, Bartsch P, Willemsen D, Oldridge N, Bjarnason-Wehrens B. Resistance and balance training improves functional capacity in very old participants attending cardiac rehabilitation after coronary bypass surgery. J Am Geriatr Soc. 2012 Dec;60(12):2270-6. doi: 10.1111/jgs.12030. Epub 2012 Nov 23. PMID 23176104
- [Background] Salavati M, Fallahinia G, Vardanjani AE, Rafiei H, Mousavi S, Torkamani M. Comparison Between Effects of Home Based Cardiac Rehabilitation Programs Versus Usual Care on the Patients' Health Related Quality of Life After Coronary Artery Bypass Graft. Glob J Health Sci. 2015 Aug 19;8(4):196-202. doi: 10.5539/gjhs.v8n4p196. PMID 26573042
- [Background] Arefi S. Phase of cardiac rehabilitation programs on anxiety and depression in patients with acute coronary syndrome. 2012.
- [Background] Sibilitz KL, Berg SK, Hansen TB, Risom SS, Rasmussen TB, Hassager C, Kober L, Gluud C, Thygesen LC, Lindschou J, Schmid JP, Taylor RS, Zwisler AD. Update to the study protocol, including statistical analysis plan for a randomized clinical trial comparing comprehensive cardiac rehabilitation after heart valve surgery with control: the CopenHeartVR trial. Trials. 2015 Feb 5;16:38. doi: 10.1186/s13063-015-0562-z. PMID 25887433
- [Background] Kang Y, Yang IS. Cardiac self-efficacy and its predictors in patients with coronary artery diseases. J Clin Nurs. 2013 Sep;22(17-18):2465-73. doi: 10.1111/jocn.12142. Epub 2013 Feb 27. PMID 23441807
- [Background] Borzou SR, Amiri S, Salavati M, Soltanian AR, Safarpoor G. Effects of the First Phase of Cardiac Rehabilitation Training on Self-Efficacy among Patients Undergoing Coronary Artery Bypass Graft Surgery. J Tehran Heart Cent. 2018 Jul;13(3):126-131. PMID 30745925
- [Background] Babu AS, Noone MS, Haneef M, Naryanan SM. Protocol-Guided Phase-1 Cardiac Rehabilitation in Patients with ST-Elevation Myocardial Infarction in A Rural Hospital. Heart Views. 2010 Jun;11(2):52-6. doi: 10.4103/1995-705X.73209. PMID 21187997
- [Background] Dalal HM, Doherty P, Taylor RS. Cardiac rehabilitation. BMJ. 2015 Sep 29;351:h5000. doi: 10.1136/bmj.h5000. No abstract available. PMID 26419744
- [Background] Evans ES. Cardiovascular and blood lactate responses to low, moderate, and high intensity aerobic exercise in breast cancer patients: Is exercise intensity a true reflection of perceived exertion? : The University of North Carolina at Chapel Hill; 2008.
- [Background] Whaley MH, Brubaker PH, Otto RM, Armstrong LE. ACSM's guidelines for exercise testing and prescription: Lippincott Williams & Wilkins; 2006.
- [Background] Thow M. Exercise leadership in cardiac rehabilitation: an evidence-based approach: John Wiley & Sons; 2006.
- [Background] De Jonghe B, Sharshar T, Lefaucheur JP, Authier FJ, Durand-Zaleski I, Boussarsar M, Cerf C, Renaud E, Mesrati F, Carlet J, Raphael JC, Outin H, Bastuji-Garin S; Groupe de Reflexion et d'Etude des Neuromyopathies en Reanimation. Paresis acquired in the intensive care unit: a prospective multicenter study. JAMA. 2002 Dec 11;288(22):2859-67. doi: 10.1001/jama.288.22.2859. PMID 12472328
- [Background] Berry MJ, Morris PE. Early exercise rehabilitation of muscle weakness in acute respiratory failure patients. Exerc Sport Sci Rev. 2013 Oct;41(4):208-15. doi: 10.1097/JES.0b013e3182a4e67c. PMID 23873130